CLINICAL TRIAL: NCT00257920
Title: A Phase 4, Single-Center, Open-Label, Randomized, Active-Controlled, Cross-over Pilot Study to Evaluate the Effects of Two Vitamin D Analogs, Zemplar® Injection and Hectorol® Injection, on Intestinal Absorption of Calcium in CKD Stage 5 Subjects on Hemodialysis
Brief Title: A Study of Zemplar® Injection and Hectorol® Injection on Intestinal Absorption of Calcium in Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Dennis Andress, MD, Senior Medical Director, Renal Global Project Team, Abbott
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M04-726
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Results first posted 2009-05-20 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Chronic Kidney Disease, Stage 5; Secondary Hyperparathyroidism
Keywords: Stage 5 Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary | interventions — paricalcitol; 1 alpha-hydroxyergocalciferol

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Zemplar® injection
- B (Active Comparator)
  Interventions: Drug: Hectorol® injection

INTERVENTIONS:
Drug: Zemplar® injection — 6 mcg QOD
  Other Names: ABT-358; paricalcitol; Zemplar
  Arms: A
Drug: Hectorol® injection — 3.6 mcg QOD
  Other Names: Hectorol®
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the effects of Zemplar® Injection and Hectorol® Injection on intestinal calcium absorption in Chronic Kidney Disease Stage 5 subjects on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >= 20 years of age.
* Subject is diagnosed with CKD Stage 5, and must be on maintenance (chronic) hemodialysis (HD) three times a week for at least 2 months prior to the Screening Visit and expected to remain on HD for the duration of the study.
* If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control:

  * Condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD)
  * Contraceptives (oral or parenteral) for three months prior to study drug administration
  * In a monogamous relationship with a vasectomized partner
* If female, subject is not breastfeeding and has a negative serum pregnancy test prior to the treatment phase.
* Subject has an intact PTH value > 200 pg/mL at Screening only (or Re-screening, if applicable).
* Subject has a serum calcium level < 10.2 mg/dL at Screening only (or Re-screening, if applicable).
* Subject has a serum phosphorus level < 6.5 mg/dL at Screening only (or Re-screening, if applicable).
* Subject has a CaxP product <= 65 at Screening only (or Re-screening, if applicable).
* Subject must voluntarily sign and date an informed consent, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to the conduct of any study-specific procedure.

Exclusion Criteria:

* Subject has a history of an allergic reaction or significant sensitivity to vitamin D or vitamin D related compounds.
* Subject has chronic gastrointestinal disease, which in the Investigator's opinion, may result in clinically significant GI malabsorption.
* Liver function defects defined as > 2 times the upper limit of normal for liver enzyme (SGOT/AST, SGPT/ALT) levels.
* Subject has a hemoglobin level < 9.0 g/dL.
* Subject is taking maintenance calcitonin, Sensipar® (cinacalcet), glucocorticoids in an equivalent dose > 5 mg prednisone daily, or other drugs that may affect calcium or bone metabolism within 2 weeks prior to screening, other than females on stable (same dose and product for 3 months) estrogen and/or progestin therapy.
* For any reason, subject is considered by the Investigator to be an unsuitable candidate to receive pharmacological doses of vitamin D.
* Subject has received any investigational drug within 4 weeks prior to the Treatment Phase.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-06; Primary Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Bellevue, Nebraska
  - Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects assigned randomly in a 1:1 manner to Sequence Group I or II. Group I received Drug A (6 mcg Zemplar Injection QOD for 6 doses) in Period 1 and Drug B (3.6 mcg Hectorol Injection QOD for 6 doses) in Period 2. Each treatment period was 14 days and a 14 day washout separated the treatment periods.
Groups:
- Zemplar First: 6 mcg Zemplar Injection every other day (QOD) for 6 doses in Period 1 and 3.6 mcg Hectorol Injection for 6 doses in Period 2
- Hectorol First: 3.6 mcg Hectorol Injection QOD for 6 doses in Period 1 and 6 mcg Zemplar Injection QOD for 6 doses in Period 2
Period: Period: First Intervention
Arm/Group | Zemplar First | Hectorol First
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0
Period: Period: Washout Period of Two Weeks
Arm/Group | Zemplar First | Hectorol First
Started | 21 | 20
Completed | 21 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Period: Second Intervention
Arm/Group | Zemplar First | Hectorol First
Started | 21 | 19
Completed | 19 | 18
Not Completed | 2 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Zemplar First: 6 mcg Zemplar Injection QOD for 6 doses in Period 1 and 3.6 mcg Hectorol Injection QOD for 6 doses in Period 2
- Total: Total of all reporting groups
Arm/Group | Zemplar First | Hectorol First | Total
Number analyzed (Participants) | 21 | 20 | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.03) | 55.6 (9.81) | 55.0 (10.34)
Age, Customized [Number; unit: participants]
  <40 years | 2 | 1 | 3
  40 - <60 years | 13 | 12 | 25
  >=60 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 15 | 7 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 15 | 33
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 0 | 0 | 0
  No ethnicity | 21 | 20 | 41
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41
Calcium Absorption Fraction [Mean (Standard Deviation); unit: Fractions] — Calcium Absorption Fraction= 5-hr calcium specific activity (fraction of oral dose per gram calcium) adjusted for body size differences
  Fractions | 0.085 (0.0086) | 0.130 (0.0132) | 0.107 (0.0085)

OUTCOME MEASURES:

1. Secondary Outcome: Calcium Absorption Fractions Analyzed by Mixed Model
Description: Calcium Absorption Fraction obtained at the end of Period 1 & Period 2
Time Frame: 42 Days
Population: ITT Population -all randomized subjects who received at least one dose of study drug and were analyzed by the randomized treatment sequence assigned to each subject.
Measure: Least Squares Mean (Standard Error); unit: Fractions
Groups:
- Zemplar: 6 mcg Zemplar Injection QOD for 6 doses in Period 1 or Period 2
- Hectorol: 3.6 mcg Hectorol Injection QOD for 6 doses in Period 1 or Period 2.
Arm/Group | Zemplar | Hectorol
Number analyzed (Participants) | 36 | 37
Fractions | 0.106 (0.011) | 0.110 (0.011)
Statistical Analysis 1: Comparison: Zemplar vs Hectorol; The null hypothesis was that there is no difference in the mean calcium absorption fraction between Zemplar Injection and Hectorol Injection. The power calculation applied to the primary efficacy analysis; Test type: Superiority or Other; p = 0.670, Mixed Models Analysis — No adjustment was made for multiple comparisons. A single hypothesis was tested by the primary efficacy analysis. All hypothesis tests were two-tailed and P-values <= 0.050 were considered statistically significant; Mean Difference (Final Values) = -0.004, 95% CI [-0.023 to 0.015], Standard Error of Mean 0.009

2. Primary Outcome: Calcium Absorption Fractions Analyzed by Analysis of Variance (ANOVA)
Description: Calcium Absorption Fraction obtained at the end of Period 1 & Period 2
Time Frame: 42 Days
Population: Per-Protocol Population - all subjects who completed both Period 1 and 2 and did not have major protocol violations.
Measure: Least Squares Mean (Standard Error); unit: Fractions
Arm/Group | Zemplar | Hectorol
Number analyzed (Participants) | 33 | 33
Fractions | 0.103 (0.007) | 0.108 (0.007)
Statistical Analysis 1: Comparison: Zemplar vs Hectorol; The null hypothesis was that there is no difference in mean calcium absorption between Zemplar and Hectorol. Approximately 42 subjects were to be randomized assuming 36 subjects would available in the per-protocol set. A sample size of 36 subjects has 80% power to detect a mean difference of -0.018 assuming the Zemplar group mean is 0.139, the Hectorol group mean is 0.157 and the STD is 0.037. The ANOVA model included effects for sequence, subject-within-sequence, period and treatment regimen; Test type: Superiority or Other; p = 0.573, ANOVA — No adjustment was made for multiple comparisons. A single hypothesis was tested by the primary efficacy analysis. All hypothesis tests were two-tailed and P-values <=0.050 were considered statistically significant; Mean Difference (Final Values) = -0.005, 95% CI [-0.024 to 0.014], Standard Error of Mean 0.009

ADVERSE EVENTS:
Groups:
- Zemplar: 6mcg Zemplar Injection QOD for 6 doses in Period 1 or Period 2.
Arm/Group | Zemplar | Hectorol
Serious Adverse Events (participants affected / at risk) | 3 | 3
Other Adverse Events (participants affected / at risk) | 18 | 15
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Zemplar | Hectorol
Hypoaesthesia (Nervous system disorders) | 1/40 (1) | 0/41 (0)
Dizziness (Nervous system disorders) | 0/40 (0) | 1/41 (1)
Arterial Stenosis (Vascular disorders) | 1/40 (1) | 0/41 (0)
Thrombosis (Vascular disorders) | 1/40 (1) | 0/41 (0)
Palpitations (Cardiac disorders) | 0/40 (0) | 1/41 (1)
Tachycardia (Cardiac disorders) | 0/40 (0) | 1/41 (1)
Diarrhoea (Gastrointestinal disorders) | 0/40 (0) | 1/41 (1)
Abdominal Pain (Gastrointestinal disorders) | 0/40 (0) | 1/41 (1)
Nausea (Gastrointestinal disorders) | 0/40 (0) | 3/41 (3)
Vomiting (Gastrointestinal disorders) | 0/40 (0) | 2/41 (2)
Anxiety (Psychiatric disorders) | 0/40 (0) | 1/41 (1)
Asthenia (General disorders) | 0/40 (0) | 1/41 (1)
Chest Pain (General disorders) | 0/40 (0) | 1/41 (1)
Fatigue (General disorders) | 0/40 (0) | 1/41 (1)
Oedema Peripheral (General disorders) | 1/40 (1) | 1/41 (1)
Suprapubic pain (General disorders) | 0/40 (0) | 1/41 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/40 (1) | 0/41 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0/40 (0) | 1/41 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/40 (0) | 1/41 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0/40 (0) | 1/41 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0/40 (0) | 1/41 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0/40 (0) | 1/41 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Zemplar | Hectorol
Constipation (Gastrointestinal disorders) | 1/40 (1) | 1/41 (1)
Nausea (Gastrointestinal disorders) | 1/40 (1) | 0/41 (0)
Vomiting (Gastrointestinal disorders) | 1/40 (1) | 0/41 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0/40 (0) | 1/41 (1)
Diarrhoea (Gastrointestinal disorders) | 1/40 (1) | 0/41 (0)
Eye infection (Infections and infestations) | 1/40 (1) | 0/41 (0)
Nasopharyngitis (Infections and infestations) | 1/40 (1) | 1/41 (1)
Fall (Injury, poisoning and procedural complications) | 1/40 (1) | 1/41 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0/40 (0) | 1/41 (1)
Hypoacusis (Ear and labyrinth disorders) | 1/40 (1) | 0/41 (0)
Diabetic retinal oedema (Eye disorders) | 0/40 (0) | 1/41 (1)
Chest pain (General disorders) | 2/40 (2) | 0/41 (0)
Chills (General disorders) | 0/40 (0) | 1/41 (1)
Local swelling (General disorders) | 1/40 (1) | 0/41 (0)
Malaise (General disorders) | 1/40 (1) | 1/41 (1)
Oedema Peripheral (General disorders) | 2/40 (2) | 0/41 (0)
Pain (General disorders) | 1/40 (1) | 1/41 (1)
Pyrexia (General disorders) | 0/40 (0) | 1/41 (1)
Bleeding time prolonged (Investigations) | 1/40 (1) | 0/41 (0)
Blood glucose decreased (Investigations) | 1/40 (1) | 1/41 (1)
Blood potassium decreased (Investigations) | 0/40 (0) | 1/41 (1)
Blood pressure increased (Investigations) | 1/40 (1) | 0/41 (0)
Body temperature increased (Investigations) | 0/40 (0) | 1/41 (1)
Cardiac murmur (Investigations) | 0/40 (0) | 1/41 (1)
Culture urine positive (Investigations) | 1/40 (1) | 0/41 (0)
Heart rate irregular (Investigations) | 1/40 (1) | 0/41 (0)
Urine output decreased (Investigations) | 0/40 (0) | 1/41 (1)
Weight decreased (Investigations) | 0/40 (0) | 1/41 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/40 (1) | 1/41 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1/40 (1) | 0/41 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2/40 (2) | 0/41 (0)
Paraesthesia (Nervous system disorders) | 1/40 (1) | 0/41 (0)
Hypoaesthesia (Nervous system disorders) | 1/40 (1) | 0/41 (0)
Insomnia (Psychiatric disorders) | 1/40 (1) | 0/41 (0)
Dysuria (Renal and urinary disorders) | 0/40 (0) | 1/41 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1/40 (1) | 2/41 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/40 (2) | 0/41 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/40 (1) | 0/41 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1/40 (1) | 0/41 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0/40 (0) | 2/41 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0/40 (0) | 1/41 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1/40 (1) | 0/41 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0/40 (0) | 1/41 (1)
Haemorrhage (Vascular disorders) | 0/40 (0) | 1/41 (1)
Thrombosis (Vascular disorders) | 1/40 (1) | 0/41 (0)

LIMITATIONS AND CAVEATS:
The null hypothesis was not tested appropriately as a result of measurable differences in parathyroid hormone (PTH) suppression indicating dose exposure was different. Therefore, differences in calcium absorption could not be determined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days